CLINICAL TRIAL: NCT05661864
Title: Multi-Tiered Systems of Teacher Training and Classroom Management
Brief Title: Multi-Tiered Systems of Support for Teacher Training in Classroom Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Kentucky University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1950299-1
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Universal Behavioral Supports; Teacher Training

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups. Both groups receive intervention, but to different classroom management strategies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Tiered Systems of Support for Teacher Training Evaluation (Experimental): Participants will be randomized to a target practice group. The group will receive the multi-tiered systems of support (online instruction, self-monitoring, self-management) for the target practice. They will not receive instruction on the non-target practice until after study data collection concludes.
  Interventions: Behavioral: Multi-Tiered Systems of Support for Teacher Training
- Control (No Intervention): Participants will not receive intervention on the non-target practice until after study data collection concludes. This practice will serve as the comparison for the group who received intervention on the practice.

INTERVENTIONS:
Behavioral: Multi-Tiered Systems of Support for Teacher Training — In tier 1 of the intervention, all participants will complete online modules on the target practice and self-monitoring. They will then self-monitor the target practice for approximately three weeks. Non-responders will receive intensified intervention (tier 2) in which they will complete an online module on self-management. They will then self-manage their use of the target practice for approximately 3 weeks. Continued non-responders will receive peer coaching on the target practice (tier 3). Responders to tiers 2-3 will move down a tier after 3 weeks of response.
  Arms: Multi-Tiered Systems of Support for Teacher Training Evaluation

SUMMARY:
The goal of this clinical trial is to test the effects of a responsive approach to training teachers to increase their use of evidence-based classroom management practices. The main question to answer is whether teachers increase their use of a target classroom management practice when they receive the intervention. All participants will receive the intervention. The target practice for which they receive intervention will be randomly assigned. Participants will submit videos of an instructional activity in their classroom 1-2 times per week over a period of 12-15 weeks. They will be asked to complete online modules on classroom management practices and to self-monitor their use of one classroom management practice. Participants may also be asked to graph their data, watch videos of themselves teaching, or implement peer coaching with a classmate or other participant. Researchers will compare the change in target classroom management practices between groups to test if the change in the group who targeted the practice is greater than the change in the group who did not target the practice.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in EDU 502 or PK-12 classroom teacher

Exclusion Criteria:

* Inability to submit video recordings of instruction for data collection and analysis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in the frequency of the target practice | Baseline, endpoint (15 weeks from start date)
  The investigators will measure the frequency of the target practice during baseline and treatment sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Kentucky University, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided